CLINICAL TRIAL: NCT04988607
Title: The Efficacy and Safety of Osimertinib Plus Bevacizumab Versus Osimertinib Monotherapy in Treatment-naïve Advanced NSCLC Patients Harbouring EGFR Exon 21 L858R Mutation: A Prospective, Multicenter, Randomized, Open Label Study (FLAIR)
Brief Title: Osimertinib Plus Bevacizumab in Untreated EGFR Exon21 L858R Mutated NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2002
Record Dates: First submitted 2021-06-20; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1, the experimental arm is osimertinib plus bevacizumab, while the control arm is osimertinib monotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osimertinib plus bevacizumab (Experimental): Osimertinib 80 mg (QD) in combination with Bevacizumab (15 mg/kg) (Q3W)
  Interventions: Drug: Osimertinib; Drug: Bevacizumab
- osimertinib (Active Comparator): All patients randomized into this will only receive Osimertinib 80mg (QD)
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — osimertinib plus bevacizumab arm is dosed at osimertinib 80 mg orally once every day combined with bevacizumab 15mg/kg by intravenous drip infusion on day 1 of a 21-day (within 3 days) cycle
  Other Names: AZD9291; Tagrisso
  Arms: osimertinib plus bevacizumab
Drug: Bevacizumab — osimertinib plus bevacizumab arm is dosed at osimertinib 80 mg orally once every day combined with bevacizumab 15mg/kg by intravenous drip infusion on day 1 of a
  Other Names: Avastin
  Arms: osimertinib plus bevacizumab
Drug: Osimertinib — Osimertinib is dosed orally at 80 mg once per day
  Other Names: AZD9291; Tagrisso
  Arms: osimertinib

SUMMARY:
This is a prospective, multicenter, randomized, open label study to investigate the efficacy and safety of osimertinib plus bevacizumab versus osimertinib montherapy in treatment-naïve recurrent or metastatic NSCLC patients harbouring EGFR exon 21 L858R mutation.

DETAILED DESCRIPTION:
Enrolled patients will be randomized 1:1, the experimental arm is osimertinib plus bevacizumab, while the control arm is osimertinib monotherapy. Osimertinib monotherapy arm is dosed at a 80 mg once per day; osimertinib plus bevacizumab arm is dosed at osimertinib 80 mg orally once every day combined with bevacizumab 15mg/kg by intravenous drip infusion on day 1 of a 21-day (within 3 days) cycle. All treatment will be done continuously until RECIST 1.1-defined progression as assessed by the Investigator or another discontinuation criterion is met.

Patients will undergo the efficacy assessments based on RECIST 1.1 assessment criterion every 6 weeks, until disease progression as assessed by the Investigator. The follow-up assessment after disease progression will be repeated every 12 weeks until study complete.

In addition, patients will undergo the safety assessment in the whole treatment period and 28-day safety follow-up after discontinued study drug for any reason or study complete.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, subjects should fulfil the following criteria based on local regulations:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
2. Provision of signed and dated, written informed consent form prior to any mandatory study-specific procedures, sampling, and analyses.
3. Male or female, age ≥18 years old.
4. Newly diagnosed metastatic NSCLC (clinical stage IVA or IVB) or recurrent NSCLC (per Version 8 of the International Association for the Study of Lung Cancer [IASLC] Staging Manual in Thoracic Oncology), not amenable to curative surgery or radiotherapy.
5. Histologically or cytologically documented non-squamous NSCLC
6. Documented EGFR exon 21 L858R mutation
7. ECOG performance status of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks
8. Life expectancy ≥12 weeks at Day 1.
9. At least 1 measurable extracranial lesion according to RECIST 1.1; (Note: ① At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter with computed tomography (CT) or magnetic resonance imaging (MRI). ② CT/MRI scan slice thickness/interval no greater than 5 mm. ③ 10 mm caliper measurement by clinical examination (lesions that cannot be accurately measured with calipers should be recorded as nonmeasurable) ④ If brain metastases were received radiotherapy, these brain metastasis can't be as target lesions).
10. Patients with CNS metastases whose condition was neurologically stable 2 weeks (after steroids treatment or non-treatment) will be allowed, including leptomeningeal metastases
11. Patients who have undergone radiotherapy may be enrolled if the participants meet the following conditions • The patient has no history of radiotherapy for lesions in lung fields within 28 days before the randomization.

    • For radiotherapy outside the chest region, at least 28 days have elapsed by the time of randomization since the final irradiation date. (if the radiotherapy given as palliation to bone metastases within 2 weeks, the patient should recovery from all toxicities)
12. Adequate haematological function:

    • Absolute neutrophil count (ANC)≥1.5×109/L* AND

    • Platelet count≥100×109/L* AND

    • Haemoglobin≥9 g/dL (may be transfused to maintain or exceed this level)

    *The use of granulocyte colony stimulating factor support and platelet transfusion to meet these criteria is not permitted.
13. Adequate liver function. • Total bilirubin<1.5×upper limit of normal (ULN) AND •Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)<2.5×ULN in patients without liver metastases; <5×ULN in patients with liver metastases
14. Adequate renal function

    •Serum creatinine≤1.5×ULN or calculated creatinine clearance≧45mL/min AND
    * Urine dipstick for proteinuria<2+. Patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate≤1 g of protein in 24 hours.
15. International normalised ratio (INR)≤1.5 and partial prothrombin time (PTT or aPTT)≤1.5×ULN within 7 days prior to randomization.
16. Female patients who are not abstinent (in line with the preferred and usual lifestyle choice of the patient) and intend to be sexually active with a male partner must be using highly effective contraceptive measures, must not be breast feeding, and must have a negative pregnancy test prior to first dose of treatment or must have evidence of non-child-bearing potential by fulfilling 1 of the following criteria at screening:

    • Post-menopausal, defined as more than 50 years of age and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.

    • Women under 50 years old would be considered as postmenopausal if the participants have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.

    • Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
17. Male subjects should be willing to agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below:

    * With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 4 months after the last dose of Osimertinib.
    * Men must refrain from donating sperm during this same period

Exclusion Criteria:

1. Spinal cord compression; symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids. Patients with asymptomatic brain metastases can be eligible for inclusion if in the opinion of the Investigator immediate definitive treatment is not indicated.
2. Past medical history of ILD, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD 3. History or evidence of inherited bleeding diathesis or coagulopathy that increases the risk of bleeding.

4. Uncontrolled hypertension (blood pressures: systolic>150 mmHg and/or diastolic >100 mmHg).

5. Prior history of hypertensive crisis or hypertensive encephalopathy. 6. Significant vascular disease (including but not limited to aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization.

7. Any of the following cardiac criteria:

• Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine-derived QTcF value;

* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG; eg, complete left bundle branch block, third-degree heart block, second-degree heart block;
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as electrolyte abnormalities including serum/plasma potassium*, magnesium* and calcium* below the lower limit of normal (LLN), heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.

  * Levels must be in the normal range prior to first administration of osimertinib.

    8. Malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent.

    9. Any unresolved toxicities from prior systemic therapy (eg, adjuvant chemotherapy) greater than CTCAE Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2 prior platinum-therapy related neuropathy.

    10. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib 11. History of haemoptysis, defined as > 2.5 ml of red blood per event within 3 months prior to randomization.

    11. History of haemoptysis, defined as > 2.5 ml of red blood per event within 3 months prior to randomization.

    12. Evidence of tumour invading major blood vessels on imaging. The investigator or the local radiologist must exclude evidence of tumour that is fully contiguous with, surrounding, or extending into the lumen of a major blood vessel (e.g., pulmonary artery or superior vena cava).

    13. Non-healing wound, active peptic ulcer, or bone fracture 14. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of enrolment.

    14. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of enrolment.

    15. History of tracheo-oesophageal fistula. 16. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active gastroduodenal ulcer disease 16. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active gastroduodenal ulcer disease.

    17. Evidence of ongoing or active infection requiring IV antibiotics; any other disease, neurological, or metabolic dysfunction; physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.

    18. Prior chemotherapy or treatment with another systemic anti-cancer agent (e.g., monoclonal antibody, tyrosine kinase inhibitors, EGFR inhibitors, VEGF receptor inhibitors) for the treatment of the patient's current stage of disease (Stage IV or postoperative recurrent disease). NOTE: i. Previous adjuvant or neo-adjuvant treatment for non-metastatic disease is permitted if completed ≥ 6 months before randomization.

    19. Previous treatment received in the present study. 20. Major surgery (including open biopsy) or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during study treatment.

    21. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device are excluded within 7 days prior to initiation of study treatment. Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.

    22. Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4 (at least 3 weeks prior).

    23. Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (325 mg/day) or other nonsteroidal anti-inflammatory agents known to inhibit platelet function.

    24. Current or recent (within 10 days of first dose of bevacizumab) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes. Prophylactic use of anticoagulants is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of osimertinib plus bevacizumab treatment compared with osimertinib monotherapy | up to 3 years after the first patient is randomized
  Progression free survival (PFS) by Investigator assessment as defined by RECIST 1.1

SECONDARY OUTCOMES:
OS rate at 24 months | the Kaplan-Meier estimate of OS at 24 months
  Proportion of patients alive at 24 months
TTime to treatment failure (TTF) | up to 3 years after the first patient is randomized
  The time from date of randomization until the date of death from any cause, or the last date of osimertinib / bevacizumab treatment, or the the date before new systemic treatment other than osimertinib or bevacizumab, whichever is earlier.
Objective Response Rate (ORR) | up to 3 years after the first patient is randomized
  The number (percent) of patients with at least 1 visit response of CR or PR (per RECIST 1.1 using Investigator assessments).
Disease Control Rate (DCR) | up to 3 years after the first patient is randomized
  The percentage of subjects who have a best overall response of CR or PR or SD by RECIST 1.1 as assessed by the Investigator
Duration of Response (DoR) | up to 3 years after the first patient is randomized
  The time from the date of first documented response until the date of documented progression or death in the absence of disease progression
Central Nervous System Progression-Free Survival (CNS PFS) | up to 3 years after the first patient is randomized
  The time from randomization until the date of objective CNS progression (as defined by RECIST1.1) or death (by any cause in absence of CNS progression) regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to CNS progression
Central Nervous System Objective Response Rate (CNS ORR) | up to 3 years after the first patient is randomized
  the percentage of patients who had at least 1 visit with CNS response of PR or CR by Investigator assessment
Central Nervous System Disease Control Rate (CNS DCR) | up to 3 years after the first patient is randomized
  The percentage of subjects who have a best CNS response of CR or PR or SD by RECIST 1.1 as assessed by the Investigator
Central Nervous System Duration of Response (CNS DoR) | up to 3 years after the first patient is randomized
  The time from the date of first documented CNS response until the date of documented CNS progression or death in the absence of CNS progression
Incidence of Adverse Event (AE) | up to 3 years after the first patient is randomized
  The incidence rate of any untoward medical occurrence in a subject or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of ≥grade 3 Adverse Event (AE) | up to 3 years after the first patient is randomized
  The incidence rate of ≥grade 3 untoward medical occurrence in a subject or clinical study subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Incidence of Adverse Drug Reactions (ADR) | up to 3 years after the first patient is randomized
  The incidence rate of Adverse Events suspected to be causally related to the medicinal product.
Incidence of Adverse Events of Special Interest (AESI) | up to 3 years after the first patient is randomized
  The incidence rate of adverse events of scientific and medical interest which require close monitoring and rapid communication by the treating physician to sponsor and AstraZeneca, including ILD/pneumonitis-like event, QTc prolongation and changes in cardiac contractility

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China